CLINICAL TRIAL: NCT01955083
Title: Analysis of Snore Sound Following Minimal Invasive Surgery in Sleep-disordered Breathing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hyli38
Record Dates: First submitted 2010-07-29; First posted 2013-10-07 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2013-10

CONDITIONS: Primary Snoring; Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; snoring; radiofrequency; pillar implant; snore sound analysis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pillar implant (Experimental): Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring.
  Interventions: Device: Pillar implant
- Radiofrequency (Active Comparator): Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring.
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Pillar implant — Subjects receive pillar implant of the soft palate under local anesthesia as an outpatient procedure on sitting position. Using the delivery tool of the pillar implant system, the mucosa of the soft palate close to the hard palate-soft palate junction (approximate 0.5 cm) was punctured in the midline. The needle was inserted to the uvular muscle and moved parallel to the curve of the soft palate towards the tip of the uvula. After reaching the insertion point, the implant was delivered steadily after which the needle was withdrawn. This process was repeated for the second and third implants in the bilateral para-midline with a 0.2 cm horizontal distance from the first implant.
  Other Names: Pillar implant (Medtronic Inc., USA)
  Arms: Pillar implant
Device: Radiofrequency — Subjects receive radiofrequency under local anesthesia as an outpatient procedure on sitting position. radiofrequency energy was delivered via a generator (Somnus® Model S2, Gyrus-ACMI Corporation, Maple Grove, MN, USA) with the power set to 10 watts and the maximal target temperature to 85°C. The needle electrode was inserted through the mucosa into the muscle layer at the entry points (approximately 1 cm below the hard palate-soft palate junction). The electrode was kept in place until 600 J had been delivered at the midline and 300 J at both para-midline sites (approximately 1 cm horizontal distance).
  Other Names: Somnus® Model S2 (Gyrus-ACMI Corporation, USA)
  Arms: Radiofrequency

SUMMARY:
1. Background：The methods of anti-snore (treatment of snoring ) can be divided into conservative, invasive and minimal invasive treatment. IN brief, minimal invasive surgery involving radiofrequency and pillar implant demonstrates significantly improvement of snoring without major complication. Previous studies usually evaluated snoring through subjective measures such as visual analog scale visual analog scale. Rare reports analyzed snore sound instrumentally and no report demonstrates the correlation between subjective perception and objective assessment of snoring before and after surgical intervention.
2. Purposes：

   1. Development of snore sound spectrum.
   2. Exploration of the correlation between subjective perception and objective assessment of snoring.
   3. Comparison of changes in snoring before and after minimal invasive surgery and between two kinds of MIS to have a understanding of surgical impact in subjective and objective measurement.
3. Method：We plan to enroll 30 subjects diagnosed by polysomnography as simple snoring or mild OSA with major complaint of snoring and favorable anatomic structure for minimal invasive surgery. All eligible subjects will be instructed the purpose, process and all related rights of this study and sign inform consent in outpatient clinic. Subjects start to complete Snore Outcome Survey (SOS, a validated questionnaire) and visual analog sure of snoring (VAS). Objective overnight snore sound recoding is arranged in sleep center. Subjects then receive minimal invasive surgery：radiofrequency or pillar implant of the soft palate by randomization. Both radiofrequency and pillar implant are common techniques in treating snoring and performed under local anesthesia as an outpatient procedure on sitting position. All subjects received repeated snore sound recording and completion of SOS and VAS three months after MIS.
4. Outcomes

   1. Development of snore sound spectrum in sleep-disorder breathing patients.
   2. Correlation of parameters between snore sound recording (loudness, frequency, count, regularity, etc ) and clinical parameters.
   3. Correlation between objective (snore sound analysis) and subjective (SOS,VAS) assessment of snoring.
   4. Comparison of changes in snoring (particular in objective assessment) after radiofrequency or pillar implant.
   5. Comparison of changes in snoring between radiofrequency and pillar implant.

DETAILED DESCRIPTION:
Recent publications have demonstrated reductions in snoring with several minimal invasive surgery (MIS) methods of the soft palate including radiofrequency (RF) surgery and pillar implant (PI). Despite modest effects in the treatment of obstructive sleep apnea, patients often wish to receive MIS for habitual snoring. However, the efficacy in reducing snoring has mainly been determined by self-reported questionnaires in the past. Further, the definition of surgical success in snoring treatment has not been universally defined. To date, changes in snoring sound characteristics following MIS have not been demonstrated.

Many cohort studies and a few randomized controlled trials or clinical controlled trials have compared MIS with a placebo, different energy generators, different material rigidity, or different operative techniques. RF of the soft palate produces volumetric tissue reduction and selective scar tissue5 to reduce obstruction and induce stiffness. However, the RF energy delivered to the soft palate can be inadequate and may result in residual or recurrent snoring. PI can decrease palatal flutter by increasing the rigidity of the soft palate through implant identity and tissue fibrosis. In addition, PI can be chronically retained in the muscle layer of the soft palate thereby producing a long-term anti-snoring effect. Nevertheless, whether PI provides a better efficacy in the treatment of snoring than RF surgery is still unknown.

The primary aim of the current study was to compare the anti-snoring effect between PI and RF by subjective assessments in a randomized controlled parallel trial. The secondary aim was to explore and compare the acoustic changes in snoring sounds after PI and RF.

ELIGIBILITY:
Inclusion Criteria:

1. simple snoring or mild obstructive sleep apnea
2. major complaint of snoring
3. favorable anatomic structure for minimal invasive surgery.

Exclusion Criteria:

1. moderate or severe obstructive sleep apnea
2. pathological obesity
3. significant craniofacial anomaly
4. elderly
5. unfavorable anatomic structure for minimal invasive surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh Yu Li, professor, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

REFERENCES:
- [Background] Lee LA, Yu JF, Lo YL, Chen NH, Fang TJ, Huang CG, Cheng WN, Li HY. Comparative effects of snoring sound between two minimally invasive surgeries in the treatment of snoring: a randomized controlled trial. PLoS One. 2014 May 9;9(5):e97186. doi: 10.1371/journal.pone.0097186. eCollection 2014. PMID 24816691
- See also: Chang Gung Memorial Hospital at Linkou is a tertiary medical center in Taiwan (R.O.C.). — http://www.cgmh.org.tw/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a prospective, randomized, parallel-controlled trial in a tertiary medical center (Department of Otorhinolaryngology, Head and Neck Surgery, Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan). Subjects were recruitment from October 1, 2010 to March 31, 2012.
Pre-assignment Details: The additional inclusion criteria were: a) length of the soft palate ≥ 2.5 cm and b) the width of the base of the uvular ≥ 1.0 cm. The exclusion criteria were: a) tonsillar hypertrophy; b) high tongue position; c) retrognathia; d) craniofacial abnormalities, e) trismus, f) allergy to anesthetic, and g) poorly controlled medical disorders.
Groups:
- Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Subjects receive radiofrequency under local anesthesia as an outpatient procedure on sitting position. radiofrequency energy was delivered via a generator (Somnus® Model S2, Gyrus-ACMI Corporation, Maple Grove, MN, USA) with the power set to 10 watts and the maximal target temperature to 85°C. The needle electrode was inserted through the mucosa into the muscle layer at the entry points (approximately 1 cm below the hard palate-soft palate junction). The electrode was kept in place until 600 J had been delivered at the midline and 300 J at both para-midline sites (approximately 1 cm horizontal distance).
- Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Subjects receive pillar implant of the soft palate under local anesthesia as an outpatient procedure on sitting position. Using the delivery tool of the pillar implant system, the mucosa of the soft palate close to the hard palate-soft palate junction (approximate 0.5 cm) was punctured in the midline. The needle was inserted to the uvular muscle and moved parallel to the curve of the soft palate towards the tip of the uvula. After reaching the insertion point, the implant was delivered steadily after which the needle was withdrawn. This process was repeated for the second and third implants in the bilateral para-midline with a 0.2 cm horizontal distance from the first implant.
Period: Overall Study
Arm/Group | Radiofrequency | Pillar Implant
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency | Pillar Implant | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.3) | 38.3 (9.7) | 36.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  Taiwan | 15 | 15 | 30
VAS [Mean (Standard Deviation); unit: units on a scale] — The participants, based on descriptions from their spouse or bed partner, were asked to estimate the severity of their snoring using a 10 cm visual analogue scale (VAS) from 0 (no snoring) to 10 (very severe snoring, bed partner leaves the room).
  units on a scale | 6.8 (2.0) | 7.9 (1.7) | 7.3 (1.9)
SOS [Mean (Standard Deviation); unit: units on a scale] — The Mandarin Chinese version of the Snore Outcomes Survey (SOS) questionnaire has been validated and repeatedly used as an outcome measure in obstructive sleep apnea patients. It was comprised of eight Likert-type items to comprehensively evaluate the duration, loudness, and frequency of snoring. The scale of the SOS was normalized from 0 (worst) to 100 (best).
  units on a scale | 40.5 (9.4) | 40.4 (8.8) | 40.5 (8.9)
Total-SI [Mean (Standard Deviation); unit: event/hour] — We calculated the snoring index (SI) of the total frequency domain (40 Hz-2,000 Hz) as 'Total-SI'.
  event/hour | 116.4 (148.6) | 116.3 (94.2) | 116.3 (122.2)
Total-Imax [Mean (Standard Deviation); unit: dB] — We calculated the maximal sound intensity (Imax) of the total frequency domain (40 Hz-2,000 Hz) as 'Total-Imax'.
  dB | 57.7 (8.2) | 70.9 (13.1) | 64.3 (12.7)
Total-Imean [Mean (Standard Deviation); unit: dB] — We calculated the mean sound intensity (Imean) of the total frequency domain (40 Hz-2,000 Hz) as 'Total-Imean'.
  dB | 47.4 (7.6) | 50.8 (5.0) | 49.1 (6.6)
Total-Fpeak [Mean (Standard Deviation); unit: Hz] — We calculated the peak sound frequency (Fpeak) of the total frequency domain (40 Hz-2,000 Hz) as 'Total-Fpeak'.
  Hz | 617.3 (603.8) | 543.3 (593.1) | 580.3 (589.3)
Total-Fmean [Mean (Standard Deviation); unit: Hz] — We calculated the mean sound frequency (Fmean) of the total frequency domain (40 Hz-2,000 Hz) as 'Total-Fmean'.
  Hz | 102.3 (30.4) | 10.4 (22.7) | 101.9 (26.4)
B1-SI [Mean (Standard Deviation); unit: event/hour] — We calculated the snoring index (SI) of the low frequency domain (40 Hz-300 Hz) as 'B1-SI'.
  event/hour | 113.3 (148.9) | 113.4 (93.5) | 113.3 (122.2)
B1-Imax [Mean (Standard Deviation); unit: dB] — We calculated the maximal sound intensity (Imax) of the low frequency domain (40 Hz-300 Hz) as 'B1-Imax'.
  dB | 53.9 (7.8) | 63.8 (9.9) | 58.9 (10.1)
B1-Imean [Mean (Standard Deviation); unit: dB] — We calculated the mean sound intensity (Imean) of the low frequency domain (40 Hz-300 Hz) as 'B1-Imean'.
  dB | 44.8 (7.5) | 47.2 (4.2) | 46.0 (6.1)
B1-Fpeak [Mean (Standard Deviation); unit: Hz] — We calculated the peak sound frequency (Fpeak) of the low frequency domain (40 Hz-300 Hz) as 'B1-Fpeak'.
  Hz | 220.7 (54.8) | 217.3 (39.2) | 219.0 (46.9)
B1-Fmean [Mean (Standard Deviation); unit: Hz] — We calculated the mean sound frequency (Fmean) of the low frequency domain (40 Hz-300 Hz) as 'B1-Fmean'.
  Hz | 101.9 (28.4) | 98.0 (24.1) | 100.0 (26.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS Score After MIS
Description: The mean change in subjective snoring severity (VAS) at 3 months after MIS was the primary outcome measurement.
Time Frame: baseline and 3 months following surgery
Population: Twenty-eight patients completed the protocol; two study cases were not available for follow-up. Fourteen patients underwent radiofrequency surgery and 14 patients received pillar implant surgery. Accordingly, we analyzed the participants who completed the study protocol.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Change in VAS Score at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Mean change (after value-before value) in VAS score at 3 months after surgery was calculated.
- Change in VAS Score at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Mean change (after value-before value) in VAS score at 3 months after surgery was calculated.
Arm/Group | Change in VAS Score at 3 Months After Radiofrequency | Change in VAS Score at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
units on a scale | -1.4 (7.2) [-2.7 to -0.1] | -3.3 (9.0) [-5.0 to -1.6]
Statistical Analysis 1: Comparison: Change in VAS Score at 3 Months After Radiofrequency vs Change in VAS Score at 3 Months After Pillar Implant; We hypothesized that pillar implant provide a better efficacy in the treatment of snoring than radiofrequency surgery. The sample size was estimated using the primary outcome effects (VAS) in two previously published studies (Friedman 2008; Fang 2004). Using a two-tailed Wilcoxon signed-rank test (normal parent distribution; effect size, 1.0; type I error, 0.05; power, 80%), we got a sample size of 11. For considering a 20% drop-out rate, we needed at least 14 participants; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 17, 95% CI 2-sided [-14.4 to 48.4], Standard Deviation 16

2. Secondary Outcome: Change in SOS Score After MIS
Description: Change in SOS score at 3 months after radiofrequency or pillar implant were calculated.
Time Frame: baseline and 3 months following surgery
Population: Twenty-eight participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Change in SOS Score at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Mean change (after value-before value) in SOS score at 3 months after surgery was calculated.
- Change in SOS Score at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Mean change (after value-before value) in SOS score at 3 months after surgery was calculated.
Arm/Group | Change in SOS Score at 3 Months After Radiofrequency | Change in SOS Score at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
units on a scale | 13.0 [7.6 to 18.3] | 22.8 [15.3 to 30.3]
Statistical Analysis 1: Comparison: Change in SOS Score at 3 Months After Radiofrequency vs Change in SOS Score at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percent Change in Total-SI After MIS
Description: Percent change ([after value-before value]/[before value]*100) in Total-SI (event/hour) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Total-SI
Groups:
- Percent Change in Total-SI at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-SI (event/hour) before and at 3 months after surgery was calculated.
- Percent Change in Total-SI at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-SI (event/hour) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in Total-SI at 3 Months After Radiofrequency | Percent Change in Total-SI at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Total-SI | -48.9 (22.1) | -5.9 (25.6)
Statistical Analysis 1: Comparison: Percent Change in Total-SI at 3 Months After Radiofrequency vs Percent Change in Total-SI at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percent Change in Total-Imax After MIS
Description: Percent change ([after value-before value]/[before value]*100) in Total-Imax (dB) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Total-Imax
Groups:
- Percent Change in Total-Imax at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Imax (dB) before and at 3 months after surgery was calculated.
- Percent Change in Total-Imax at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Imax (dB) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in Total-Imax at 3 Months After Radiofrequency | Percent Change in Total-Imax at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Total-Imax | 11.3 (3.8) | -6.8 (5.9)
Statistical Analysis 1: Comparison: Percent Change in Total-Imax at 3 Months After Radiofrequency vs Percent Change in Total-Imax at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percent Change in Total-Imean After MIS
Description: Percent change ([after value-before value]/[before value]*100) in Total-Imean (dB) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Total-Imean
Groups:
- Percent Change in Total-Imean at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Imean (dB) before and at 3 months after surgery was calculated.
- Percent Change in Total-Imean at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Imean (dB) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in Total-Imean at 3 Months After Radiofrequency | Percent Change in Total-Imean at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Total-Imean | 18.2 (6.1) | -0.4 (5.6)
Statistical Analysis 1: Comparison: Percent Change in Total-Imean at 3 Months After Radiofrequency vs Percent Change in Total-Imean at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percent Change in Total-Fpeak After MIS
Description: Percent change ([after value-before value]/[before value]*100) in Total-Fpeak (Hz) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Total-Fpeak
Groups:
- Percent Change in Total-Fpeak at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Fpeak (Hz) before and at 3 months after surgery was calculated.
- Percent Change in Total-Fpeak at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Fpeak (Hz) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in Total-Fpeak at 3 Months After Radiofrequency | Percent Change in Total-Fpeak at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Total-Fpeak | -12.1 (26.2) | -6 (24.2)
Statistical Analysis 1: Comparison: Percent Change in Total-Fpeak at 3 Months After Radiofrequency vs Percent Change in Total-Fpeak at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Change in Total-Fmean After MIS
Description: Percent change ([after value-before value]/[before value]*100) in Total-Fmean (Hz) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Total-Fmean
Groups:
- Percent Change in Total-Fmean at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Fmean (Hz) before and at 3 months after surgery was calculated.
- Percent Change in Total-Fmean at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in Total-Fmean (Hz) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in Total-Fmean at 3 Months After Radiofrequency | Percent Change in Total-Fmean at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Total-Fmean | -10.9 (11.6) | -0.9 (8.7)
Statistical Analysis 1: Comparison: Percent Change in Total-Fmean at 3 Months After Radiofrequency vs Percent Change in Total-Fmean at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percent Change in B1-SI After MIS
Description: Percent change ([after value-before value]/[before value]*100) in B1-SI (event/hour) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of B1-SI
Groups:
- Percent Change in B1-SI at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-SI (event/hour) before and at 3 months after surgery was calculated.
- Percent Change in B1-SI at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-SI (event/hour) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in B1-SI at 3 Months After Radiofrequency | Percent Change in B1-SI at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of B1-SI | -51.8 (22.5) | -1.7 (29.5)
Statistical Analysis 1: Comparison: Percent Change in B1-SI at 3 Months After Radiofrequency vs Percent Change in B1-SI at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Percent Change in B1-Imax After MIS
Description: Percent change ([after value-before value]/[before value]*100) in B1-Imax (dB) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of B1-Imax
Groups:
- Percent Change in B1-Imax at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Imax (dB) before and at 3 months after surgery was calculated.
- Percent Change in B1-Imax at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Imax (dB) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in B1-Imax at 3 Months After Radiofrequency | Percent Change in B1-Imax at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of B1-Imax | 5.6 (3.1) | -9.4 (5.6)
Statistical Analysis 1: Comparison: Percent Change in B1-Imax at 3 Months After Radiofrequency vs Percent Change in B1-Imax at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percent Change in B1-Imean After MIS
Description: Percent change ([after value-before value]/[before value]*100) in B1-Imean (dB) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of B1-Imean
Groups:
- Percent Change in B1-Imean at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Imean (dB) before and at 3 months after surgery was calculated.
- Percent Change in B1-Imean at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Imean (dB) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in B1-Imean at 3 Months After Radiofrequency | Percent Change in B1-Imean at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of B1-Imean | 14.7 (5.5) | -4.6 (5.3)
Statistical Analysis 1: Comparison: Percent Change in B1-Imean at 3 Months After Radiofrequency vs Percent Change in B1-Imean at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percent Change in B1-Fpeak After MIS
Description: Percent change ([after value-before value]/[before value]*100) in B1-Fpeak (Hz) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of B1-Fpeak
Groups:
- Percent Change in B1-Fpeak at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Fpeak (Hz) before and at 3 months after surgery was calculated.
- Percent Change in B1-Fpeak at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Fpeak (Hz) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in B1-Fpeak at 3 Months After Radiofrequency | Percent Change in B1-Fpeak at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of B1-Fpeak | -33.5 (11.4) | -10.9 (7.9)
Statistical Analysis 1: Comparison: Percent Change in B1-Fpeak at 3 Months After Radiofrequency vs Percent Change in B1-Fpeak at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Percent Change in B1-Fmean After MIS
Description: Percent change ([after value-before value]/[before value]*100) in B1-Fmean (Hz) before and at 3 months after surgery was calculated.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of B1-Fmean
Groups:
- Percent Change in B1-Fmean at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Fmean (Hz) before and at 3 months after surgery was calculated.
- Percent Change in B1-Fmean at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percent change ([after value-before value]/[before value]*100) in B1-Fmean (Hz) before and at 3 months after surgery was calculated.
Arm/Group | Percent Change in B1-Fmean at 3 Months After Radiofrequency | Percent Change in B1-Fmean at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of B1-Fmean | -24.8 (8.7) | -1.6 (8.4)
Statistical Analysis 1: Comparison: Percent Change in B1-Fmean at 3 Months After Radiofrequency vs Percent Change in B1-Fmean at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

13. Post Hoc Outcome: Percentage of Good Response After MIS
Description: Postoperative 'VAS <=3' was traditionally defined as 'major response'. For a comprehensive profile of the outcomes, we further created another definition of 'fine response': 'postoperative VAS <=5 plus SOS >=60' post hoc in the present study. Accordingly, patients with a postoperative VAS <=3 or postoperative VAS <=5 plus SOS >=60' group was considered to have a 'good response'. Therefore, we calculated the 'good response' rate in the radiofrequency and pillar implant groups.
Time Frame: baseline and 3 months following surgery
Population: A total of 28 participants completed the follow-up protocol and two participants dropped out after surgery.
Measure: Mean (Standard Error); unit: percentage of Good Response
Groups:
- Percentage of Good Response at 3 Months After Radiofrequency: Arm 2- Radiofrequency (control group):
  15 subjects undergo radiofrequency of the soft palate for the treatment of snoring. Percentage of good response was calculated.
- Percentage of Good Response at 3 Months After Pillar Implant: Arm 1- Pillar implant (Study group):
  15 subjects undergo pillar implant surgery of the soft palate for the treatment of snoring. Percentage of good response at 3 months after surgery was calculated.
Arm/Group | Percentage of Good Response at 3 Months After Radiofrequency | Percentage of Good Response at 3 Months After Pillar Implant
Number analyzed (Participants) | 14 | 14
percentage of Good Response | 29 (12.5) | 71 (12.5)
Statistical Analysis 1: Comparison: Percentage of Good Response at 3 Months After Radiofrequency vs Percentage of Good Response at 3 Months After Pillar Implant; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected in 3 months.
Description: No known serious adverse event had been reported to our literature review. Other adverse events of radiofrequency surgery were mucosal ulcers and breakdown. Known other adverse event of pillar implant was protrusion of implant.
Arm/Group | Radiofrequency | Pillar Implant
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The major limitations to this study were unbalanced randomization in Total-Imax despite insignificant differences in other baseline parameters between the two groups and the small sample size of the study limited the subgroup analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No